CLINICAL TRIAL: NCT02844322
Title: The Efficacy of Cyclophosphamide Plus Dexamethasone Combinated With Rituximab or Bortezomib for the Newly Diagnosed Waldenström Macroglobulinemia - a Prospective Multicentre Randomized Control Trial From China
Brief Title: The Comparison of RCD Versus BCD in Newly Diagnosed Waldenström Macroglobulinemia
Acronym: BDH-WM01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015005
Record Dates: First submitted 2016-07-17; First posted 2016-07-26 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-03

CONDITIONS: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bortezomib (Experimental): Patients in this group will receive bortezomib+ cyclophosphamide+ dexamethasone as introduction chemotherapy regimen. Chemotherapeutic response will be evaluated after 3 cycles. If a MR or better response achieves, addition 3 cycles will be given. If not, patients will cross to RCD group for another 3 cycles. If a MR or better response comes out, addition 3 cycles will be given, otherwise, the patient will quit this study.
  Interventions: Drug: Bortezomib
- rituximab (Experimental): Patients in this group will receive rituximab+cyclophosphamide+ dexamethasone as introduction chemotherapy regimen. Chemotherapeutic response will be evaluated after 3 cycles. If a MR or better response achieves, addition 3 cycles will be given. If not, patients will cross to BCD group for another 3 cycles. If a MR or better response comes out, addition 3 cycles will be given, otherwise, the patient will quit this study.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib — compare the efficiency of bortezomib and rituximab in Waldenström macroglobulinemia
  Other Names: velcade
  Arms: Bortezomib
Drug: Rituximab — compare the efficiency of bortezomib and rituximab in Waldenström macroglobulinemia
  Other Names: Mabthera
  Arms: rituximab

SUMMARY:
The purpose of this study is to compare the efficacy of cyclophosphamide plus dexamethasone combined with rituximab or bortezomib regimens in newly diagnosed Waldenström macroglobulinemia patients.

DETAILED DESCRIPTION:
Newly diagnosed WM patients will be randomly assigned to BCD or RCD group for introduction chemotherapy. Chemotherapeutic response will be evaluated after 3 cycles. If a PR or better response achieves, addition 3 cycles will be given. If not, patients will be crossed to control group for another 3 cycles. If a PR or better response comes out, addition 3 cycles will be given, otherwise, the patients will quit this study.

ELIGIBILITY:
Inclusion Criteria:

1. aged >=18 years
2. diagnosed with LPL/WM
3. untreated or mild treated without standard regimens,especially untreated with rituximab and/or bortezomib
4. symptom patients
5. with life-expectancy more than 3 months.

Exclusion Criteria:

1. diagnosed with other malignancies outside B-NHL within one year(including active center neural system lymphoma)
2. transformed lymphoma
3. liver or renal function lesion unrelated to lymphoma
4. serious complications such as uncontrolled diabetes,gastric ulcer or other serious angiocardiopathy determined by the physician
5. HIV positive or active HBV infection or other uncontrolled systematic infection
6. clinical central nervous dysfunction
7. serious surgery within 30 days
8. pregnancy or baby nursing period or un-contracepted child-bearing period woman; 9. allergy to the trail drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
progress-free survival | up to 36 months

SECONDARY OUTCOMES:
Overall response rate | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doc, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Shuhua Yi, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
we will make the data publicly available according to the local law

REFERENCES:
- [Derived] Xiong W, Lyu R, Yu Y, Wang T, Yan Y, Wang Y, Liu W, An G, Deng S, Xu Y, Sui W, Huang W, Zou D, Wang J, Qiu L, Yi S. Rituximab plus cyclophosphamide and dexamethasone versus bortezomib plus cyclophosphamide and dexamethasone in newly diagnosed symptomatic Waldenstrom macroglobulinemia: a randomized controlled trial. Haematologica. 2024 May 1;109(5):1614-1618. doi: 10.3324/haematol.2023.284588. No abstract available. PMID 38205507